CLINICAL TRIAL: NCT00078611
Title: A Phase III, Multicenter, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Intravenous Antegren(TM) (Natalizumab) in Subjects With Moderately to Severely Active Crohn's Disease With Elevated C-Reactive Protein
Brief Title: A Clinical Trial of Natalizumab in Individuals With Moderately to Severely Active Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ELN100226-CD307
Record Dates: First submitted 2004-03-01; First posted 2004-03-08 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Inflammatory Bowel Disease; IBD; Gastroenterology; Regional Enteritis; Colitis
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Colitis | interventions — Natalizumab

INTERVENTIONS:
Drug: natalizumab
  Other Names: Antegren

SUMMARY:
The purpose of this trial is to evaluate natalizumab in individuals with moderately to severely active Crohn's Disease.

DETAILED DESCRIPTION:
Natalizumab is a humanized monoclonal antibody currently being investigated as a potential treatment for Crohn's disease. It is believed to work by preventing white blood cells from moving from the blood stream into the bowel tissue. These cells are thought to cause damage to the bowel, leading to the symptoms of Crohn's disease. Elan Pharmaceuticals is currently sponsoring an international study evaluating the safety and efficacy of natalizumab in individuals with moderately to severely active Crohn's disease. Individuals with Crohn's disease will be randomly assigned to receive either placebo (an inactive solution) or natalizumab by intravenous infusion (this means putting it directly into a vein in the arm). There will be a one out of two chance of receiving natalizumab and a one out of two chance of receiving placebo. Participants in the study will receive several infusions of natalizumab or placebo at 4-week intervals. Eligible participants will then have the opportunity to enroll into an extension study that will allow all participants to receive natalizumab. For those patients who do not enroll into the extension study, the total participation in this study will last for approximately 22 weeks.

ELIGIBILITY:
* Males and females 18 years of age or older
* Diagnosis of Crohn's disease for at least 6 months
* Females must not be pregnant or breastfeeding
* Must not have previously taken natalizumab
* Use of some other Crohn's disease medications is permitted, but will be closely supervised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462
Dates: Start 2004-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (75):
- United States (63):
  - Harmony Clinical Research, Oro Valley, Arizona
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Digestive Diseases Foundation, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Division of Digestive Diseases, Los Angeles, California
  - Community Clinical Trials, Orange, California
  - UCSF / Mt. Zion IBD Center, San Francisco, California
  - Shared Medical Research Foundation, Tarzana, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Rocky Mountain Gastroenterology, Golden, Colorado
  - Arapahoe Gastroenterology, Littleton, Colorado
  - Center for Medical Research, LLC, Manchester, Connecticut
  - Morowitz, Marion, Laessing, Shocket, Bashir, Steinberg, Salcedo, Washington D.C., District of Columbia
  - Malcolm Randall VA Medical Center, Gainesville, Florida
  - Borland Groover Clinic, Jacksonville, Florida
  - Miami Research Associates, Inc., Miami, Florida
  - Waterside Clinical Research Services, Inc., West Palm Beach, Florida
  - Shafran Gastroenterology Center, Winterpark, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - Outpatient Clinical Research Facility, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Drug Research Service, Inc., Metairie, Louisiana
  - Metropolitan Gastroenterology Group, PC / Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - New York Center for Clinical Research, Lake Success, New York
  - Mount Sinai School of Medicine, New York, New York
  - Rochester Institute for Digestive Diseases and Sciences, Inc., Rochester, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC., Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Inc., Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oklahoma Gastroenterology Associates, Tulsa, Oklahoma
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny Center for Digestive Health, Pittsburgh, Pennsylvania
  - Gastroenterology Associates, Providence, Rhode Island
  - Medical University of South Carolina - Digestive Disease Center, Charleston, South Carolina
  - Southeastern Clinical Research, Chattanooga, Tennessee
  - Gastroenterology Center of the Midsouth, P.C., Memphis, Tennessee
  - Summit Research Solutions, Memphis, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Austin Gastroenterology, PA, Austin, Texas
  - Atilla Ertan, MD, PA, Houston, Texas
  - Gastroenterology Clinic of San Antonio, P.A., San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - UVA Health System, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Internal Medicine Associates, Danville, Virginia
  - McGuire DVAMC GI (111N), Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Tacoma Digestive Disease Research Center, Tacoma, Washington
  - Aurora Helath Care, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (12):
  - University of Calgary, Calgary, Alberta
  - GI Research, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Liver and Intestinal Research Centre, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Health Sciences Center, Winnipeg, Manitoba
  - Queen Elizabeth II Science Center, Halifax, Nova Scotia
  - McMaster University Medical Centre, Hamilton, Ontario
  - Sunnybrook & Women's College Health Sciences Center, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Chauq Hopital Du St. Sacrement, Québec, Quebec